CLINICAL TRIAL: NCT05367167
Title: The Effect of Fibromyalgia Syndrome Accompanying Obstructive Sleep Apnea Syndrome on Clinical Findings
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, Principal Investigator, Kirsehir Ahi Evran Universitesi
Other Study IDs: 3
Record Dates: First submitted 2022-04-08; First posted 2022-05-10 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Obstructive Sleep Apnea; Fibromyalgia
Keywords: Polysomnography; Obstructive Sleep Apnea; Fibromiyalgia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Fibromyalgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients who meet the 2010 American College of Rheumatology diagnostic criteria and were diagnosed with OSAS in the sleep laboratory will be considered as the case group.
- Control group: Patients who did not meet the 2010 American College of Rheumatology diagnostic criteria and were diagnosed with OSAS in the sleep laboratory will be considered as the control group.

SUMMARY:
Fibromyalgia Syndrome (FMS) is a chronic disease that lasts for at least three months and is characterized by various symptoms such as tender points, widespread pain in the musculoskeletal system, sleep disturbance and fatigue. Obstructive sleep apnea (OSAS) is a disease characterized by repeated upper airway obstruction during sleep. Sleep disorders negatively affect the lives of individuals. The prevalence of OSAS is between 1-5% in studies and it is more common in men than in women. Fatigue, anxiety, depression and sleep disturbance are also common in patients with fibromyalgia. Likewise, the presence of symptoms such as musculoskeletal pain in patients with OSAS suggests that these two diseases may be related to each other. We planned this study to show the relationship between OSAS and fibromyalgia (FM).

DETAILED DESCRIPTION:
Our research will be carried out on patients diagnosed with OSAS after being evaluated in the sleep laboratory of the Research Hospital Department of Chest Diseases. Fibromyalgia screening will be performed on participants who are diagnosed with OSAS and accepted to participate in the study. Patients with FM according to the 2010 American College of Rheumatology diagnostic criteria will be divided into two groups as FM patients (case group) and patients who do not meet these criteria (control group). Sleep laboratory results and demographic data of all patients will be recorded. In addition, anxiety, depression and fatigue levels will be evaluated with scales. Fibromyalgia impact questionnaire will be applied to fibromyalgia patients. Our study is a cross-sectional prospective case-control study. It is not a treatment research, an interventional application will not be made to the patients.

Our hypothesis is that OSAS patients with FMS may have more fatigue, anxiety, depression, lower algometer values, and more severe OSAS findings in polysomnographic data.

ELIGIBILITY:
Inclusion Criteria:

1.18-60 years old 2. Diagnosed with OSAS in sleep laboratory examinations 3. Agree to participate in the study

Exclusion Criteria:

1. Pregnancy
2. Neuropsychiatric disease
3. Inflammatory Rheumatic Diseases
4. Morbid obesity
5. Using a device with a previous diagnosis of OSAS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Our research will be carried out in patients diagnosed with OSAS after being evaluated in the sleep laboratory of the Kırşehir EAH Department of Chest Diseases. Fibromyalgia screening will be performed on participants who are diagnosed with OSAS and accepted to participate in the study. Patients who were diagnosed with FM according to the 2010 American College of Rheumatology diagnostic criteria will be divided into two groups as FM patients (case group) and patients who do not meet these criteria will be divided into two groups as FM (control group).
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 0 day (baseline)
  "Fatigue Severity Scale" was used to evaluate the fatigue level of the participants. This scale consists of a 7-point Likert scale. 1 point means strongly disagree, 7 means strongly agree. High scores are associated with increased fatigue. Evaluates the effects of fatigue on physical function, motivation, family and social life. Turkish validity and reliability was established.
Fibromyalgia Impact Scale | 0 day (baseline)
  The fibromyalgia levels of the participants will be evaluated with the Fibromyalgia Impact Scale. High scores indicate increased disease activity. Consists of 10 questions Maximum score is 80. Turkish validity and reliability was done
Beck Anxiety and Depression Inventory. | 0 day (baseline)
  Anxiety and depression levels will be evaluated with the Beck Anxiety and Depression Inventory. Turkish validity and reliability were done.Beck Depression Inventory (BDI) is a 21-item self-assessment scale that measures characteristic attitudes and symptoms of depression. The application takes about 10 minutes to complete. It is designed for people aged 13 and over. High scores report an increased level of depression.Beck anxiety scale This test, which consists of 21 optional questions, is accepted as an internationally valid tool used to measure the severity of anxiety in individuals.Each item marked on the Beck anxiety scale has a score. None is 0 points, mild 1 point, moderate 2 points, and severe 3 points. In this way, these scores are summed after 21 questions are marked. High scores indicate an increased level of anxiety.
visual analog scale | 0 day (baseline)
  Pain levels will be evaluated with a visual analog scale. The VAS is a scale that evaluates the severity of pain with the Likert scale. Increased scores indicate severe pain.
Algometer. | 0 day (baseline)
  The pain threshold of all patients will be measured with an algometer. Measurement with an algometer is not an invasive measurement method. It shows the patient's pain sensitivity numerically according to the applied pressure.
Demografic Datas | 0 day (baseline)
  Sex, chronic disease, smoking
BMI | 0 day (baseline)
  64 / 5.000 Çeviri sonuçları Body mass index will be calculated by measuring height (cm), weight (kg),
Polisomnografi - SLEEP LATENCE | 0 day (baseline)
  Sleep latency time will be measured in polysomnography
Polisomnografi -SLEEP ACTIVITY | 0 day (baseline)
  Sleep efficiency will be measured during polysomnography
Polisomnografi -REM time | 0 day (baseline)
  REM time will be measured in minutes during polysomnography
Polisomnografi -NREM STAGES | 0 day (baseline)
  During polysomnography, NREM stages will be measured at 1 min, 2 min, and 3 min.
Polisomnografi - NUMBERS OF APNE | 0 day (baseline)
  Numbers of apnea will be recorded in polysomnographic measurements.
Polisomnografi -NUMBER OF HYPOPNEA | 0 day (baseline)
  Numbers of hypopnea will be recorded in polysomnographic measurements.
Polisomnografi -Apnea hypopnea index (AHI) REM, NONREM in polysomnography; Apnea hypopnea index (AHI) will be evaluated on a supine, non-supine basis. | 0 day (baseline)
  Apnea hypopnea index (AHI) will be evaluated as REM, NONREM, Supine, non-supine in polysomnography.According to the AHI level; It will be classified as SIMPLE SNORING (AHİ<5), LIGHT OSAS (AHİ 5-15), MEDIUM OSAS (AHİ 15-30), HEAVY OSAS (AHİ 30+ )
Polisomnografi -OXYGEN DESATURATION INDEX | 0 day (baseline)
  Minimum oxygen saturation and average oxygen saturation will be measured in polysomnography.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Asisst Prof, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Ahi Evran University, Kırşehir, City Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meresh ES, Artin H, Joyce C, Birch S, Daniels D, Owens JH, La Rosa AJ, Rao MS, Halaris A. Obstructive sleep apnea co-morbidity in patients with fibromyalgia: a single-center retrospective analysis and literature review. Open Access Rheumatol. 2019 Apr 29;11:103-109. doi: 10.2147/OARRR.S196576. eCollection 2019. PMID 31118843
- [Background] Koseoglu HI, Inanir A, Kanbay A, Okan S, Demir O, Cecen O, Inanir S. Is There a Link Between Obstructive Sleep Apnea Syndrome and Fibromyalgia Syndrome? Turk Thorac J. 2017 Apr;18(2):40-46. doi: 10.5152/TurkThoracJ.2017.16036. Epub 2017 May 1. PMID 29404158
- [Background] Mutlu P, Zateri C, Zohra A, Ozerdogan O, Mirici AN. Prevalence of obstructive sleep apnea in female patients with fibromyalgia. Saudi Med J. 2020 Jul;41(7):740-745. doi: 10.15537/smj.2020.7.25165. PMID 32601643
- [Derived] Cigdem Karacay B, Sahbaz T, Zerman N, Tuncay F. The impact of fibromyalgia syndrome on obstructive sleep apnea syndrome in terms of pain threshold, daytime symptoms, anxiety, depression, disease severity, and sleep quality: a polysomnographic study. Sleep Breath. 2023 Aug;27(4):1473-1479. doi: 10.1007/s11325-023-02831-2. Epub 2023 Apr 18. PMID 37071285